CLINICAL TRIAL: NCT04380961
Title: Phase 2, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Sirukumab in Confirmed Severe or Critical COVID-19 Disease
Brief Title: A Study to Evaluate the Efficacy and Safety of Sirukumab in Confirmed Severe or Critical Confirmed Coronavirus Disease (COVID)-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Pharmaceutica N.V., Belgium (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CR108820; CNTO136COV2001 (Other: Janssen Pharmaceutica N.V., Belgium); 2020-003056-32 (EudraCT Number)
Record Dates: First submitted 2020-05-07; First posted 2020-05-08 (Actual); Results first posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-05

CONDITIONS: Critical Confirmed Coronavirus Disease (COVID)-19
MeSH Terms: conditions — COVID-19 | interventions — sirukumab; Standard of Care

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sirukumab (Experimental): Participants will receive single intravenously (IV) dose infusion of sirukumab on Day 1 along with standard of care treatment.
  Interventions: Drug: Sirukumab; Other: Standard of Care (SOC)
- Placebo (Placebo Comparator): Participants will receive IV single dose infusion of placebo on Day 1 along with standard of care treatment.
  Interventions: Drug: Placebo; Other: Standard of Care (SOC)

INTERVENTIONS:
Drug: Sirukumab — Participants will receive single dose infusion of sirukumab on Day 1.
  Other Names: CNTO136
  Arms: Sirukumab
Drug: Placebo — Participants will receive placebo IV single dose infusion on Day 1.
  Arms: Placebo
Other: Standard of Care (SOC) — SOC treatment will be determined by the investigator based on local practice and consists of supportive care.

SUMMARY:
The purpose of this study is to evaluate the clinical response of sirukumab (administered as a single intravenous dose) plus standard of care (SOC) compared to placebo plus SOC in COVID-19.

DETAILED DESCRIPTION:
Severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2), the causative agent of coronavirus disease 2019 (COVID-19), is an enveloped, positive-sense, single-stranded ribonucleic acid (RNA) betacoronavirus. Symptoms of COVID-19 infection may appear from 2 to 14 days following exposure, with the spectrum of illnesses ranging from mild symptoms to severe illness or death. The identification of SARS-CoV-2 follows the emergence of 2 other novel betacoronaviruses: SARS-CoV and Middle East respiratory syndrome coronavirus (MERS-CoV). Current management of COVID-19 is supportive, and respiratory failure from acute respiratory distress syndrome (ARDS) is the leading cause of mortality. While an understanding of the epidemiology and clinical spectrum of COVID-19 is still evolving during the ongoing pandemic, the current knowledge of the disease burden highlights the urgent medical need to develop a treatment. Sirukumab (also known as CNTO136) is a human anti-interleukin (IL)-6 immunoglobulin G1 kappa (IgG1k) monoclonal antibody (mAb). Sirukumab binds with high affinity and specificity to human IL-6 and as a result inhibits IL-6-mediated signaling and the biological effects of IL-6. The study will include a Screening Phase (up to 1 Day), a Treatment Phase (Day 1 to Day 28) and a Follow-up Phase (post Day 28, follow-up phone calls on Week 8, Week 12 and Week 16). Safety evaluations will include monitoring of adverse events and serious adverse events, physical examinations, vital sign measurements, electrocardiograms, clinical laboratory tests, pregnancy testing, and checking of vital status. The entire study duration for each participant will be 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized
* Has laboratory-confirmed severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection as determined by real time-polymerase chain reaction (PCR) at any time before randomization
* Evidence of infiltrates by chest X-ray, chest computed tomography (CT), lung ultrasound, or chest auscultation (rales, crackles)
* Informed consent must be obtained from the participant indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study
* Critical COVID-19 disease, defined as: Requires supplemental oxygen delivered by nonrebreather mask or high-flow nasal cannula or use of non-invasive or invasive ventilation or requiring treatment in an intensive care unit

  1. AND corresponding to category 4 on the 6-point ordinal recovery scale, that is: requires one of the above modalities to sustain a peripheral capillary oxygen saturation (SpO2) greater than (>) 93 percent (%) with a fraction of inspired oxygen (FiO2) of 50% or higher. Note, the use of other devices may fit with category 4 if the FiO2 is 50% or higher.
  2. OR, corresponding to category 5 on the 6-point ordinal recovery scale, that is partial pressure of oxygen in arterial per percentage of inspired oxygen (PaO2/FiO2) ratio < 300 millimeter of mercury (mmHg) while on invasive mechanical ventilation or veno-venous extracorporeal membrane oxygenation (ECMO) for less than 48 hours prior to screening

Exclusion Criteria:

* On invasive mechanical ventilation or on veno-venous ECMO for >48 hours at time of screening
* Received an investigational intervention (including investigational vaccines) or used an invasive investigational medical device within 30 days before the planned dose of study intervention. Note: the investigator must ensure that the participant is not enrolled in another COVID-19 study with an investigational intervention (apart from the exception specified below) prior to completion of Day 28 of the current study. Exception: participation in a single arm study, a non-blinded controlled study, expanded access, compassionate use program or any other program that is not a blinded study is allowed if it is conducted with one of the following: agents with demonstrated in vitro-effect against SARSCoV- 2, as mentioned in the center of disease control and prevention (CDC) guidelines and convalescent plasma
* Current confirmed or high suspicion for pulmonary embolus, hemodynamic significant pericardial effusion, myocarditis, or Class 3 or 4 congestive heart failure as defined by the New York Heart Association Functional Classification AND/OR Current evidence of active cardiac ischemia
* Has a history of respiratory condition (that is, asthma, chronic obstructive pulmonary disease (COPD), cystic fibrosis, fibrotic lung disease) that requires home oxygen supplementation, supportive non-invasive ventilation or, is status/post lung volume reduction surgery (LVRS). Exception: Participants with sleep apnea using supportive non-invasive ventilation (continuous positive airway pressure [CPAP]) at screening may be included
* On renal replacement therapy (defined as peritoneal dialysis or hemodialysis)
* Screening laboratory test result as follows: absolute neutrophil count (ANC) <1.0*10^3 cells/microliter; Platelet count <50*10^3 cells/microliter; estimated glomerular filtration rate (eGFR) <=30 milliliter per minute per 1.73 square meter (mL/min/1.73 m^2); Bilirubin >2* upper limit of normal (ULN) unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin; alanine aminotransferase/ aspartate aminotransferase (ALT) >5*ULN; Prothrombin time (PT)/international normalized ratio (INR) >1.5*ULN or activated partial thromboplastin time (aPTT) >1.5*ULN related to known coagulopathy or bleeding disorder (the participant can receive anticoagulant therapies for underlying conditions, or as systematic thromboprophylaxis due to COVID-19, or as part of the treatment of complications of COVID-19, but cannot participate in a clinical study with anticoagulants for COVID-19)
* Pregnant or breastfeeding, unless in the opinion of the investigator, the benefit outweighs the risks
* Has active hepatitis B or C infection or has human immunodeficiency virus infection or acquired immune deficiency syndrome (HIV/AIDS) based on medical history and/or concomitant medication
* Known active or latent tuberculosis (TB), history of incompletely treated TB, suspected or known extrapulmonary TB based on medical history and/or concomitant medication
* Evidence of active bacterial (including but not limited to bacterial pneumonia), fungal, viral or opportunistic infection (other than SARS-CoV-2)
* Currently active clinically significant (example, causing hemodynamic instability and/or causing hypoxemia) and uncontrolled arrhythmia

Ages: 18 Years to 84 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2020-04-24 (Actual); Primary Completion 2021-04-09 (Actual); Study Completion 2021-06-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutica N.V., Belgium Clinical Trial, Study Director — Janssen Pharmaceutica N.V., Belgium
Locations (16):
- United States (16):
  - MemorialCare Research Miller Children's and Women's Hospital Long Beach, Long Beach, California
  - Hoag Memorial Hospital, Newport Beach, California
  - Holy Cross Hospital - Michael and Dianne Bienes Comprehensive Cancer Center, Fort Lauderdale, Florida
  - Great Lakes Clinical Trials, Chicago, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Illinois College of Medicine at Peoria, Peoria, Illinois
  - Louisiana State University Health Sciences Center, New Orleans, Louisiana
  - Henry Ford Hospital, Detroit, Michigan
  - Beaumont Health Systems, Royal Oak, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - Saint Michaels Medical Center - Infectious Disease, Newark, New Jersey
  - SUNY Upstate Medical University, Syracuse, New York
  - East Carolina University, Greenville, North Carolina
  - Baylor Scott & White Research Institute, Dallas, Texas
  - Baylor All Saints Medical Center at Fort Worth, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency.
  As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Thys K, Loza MJ, Lynn L, Callewaert K, Varma L, Crabbe M, Van Wesenbeeck L, Van Landuyt E, De Meyer S, Aerssens J, Verbrugge I. Pharmacodynamic, prognostic, and predictive biomarkers in severe and critical COVID-19 patients treated with sirukumab. Sci Rep. 2024 Oct 3;14(1):22981. doi: 10.1038/s41598-024-74196-9. PMID 39362933

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 212 participants who started the study and got randomized, 209 participants (139 in Sirukumab + Standard of Care [SOC] and 70 in Placebo + SOC arm) were treated. Out of 212, 139 participants (96 in Sirukumab + SOC and 43 in Placebo + SOC arms) completed the study.
Groups:
- Sirukumab + SOC: Hospitalized participants with confirmed severe or critical coronavirus disease-2019 (COVID-19) received intravenous (IV) single dose infusion of sirukumab (5 milligrams per kilogram [mg/kg]) on Day 1 along with standard of care (SOC) treatment per the discretion of the Investigator.
- Placebo + SOC: Hospitalized participants with confirmed severe or critical COVID-19 disease received IV single dose infusion of placebo on Day 1 along with SOC treatment per the discretion of the Investigator.
Period: Overall Study
Arm/Group | Sirukumab + SOC | Placebo + SOC
Started | 140 | 72
Treated | 139 | 70
Participants Who Entered the Follow-up Phase | 118 | 57
Completed | 96 | 43
Not Completed | 44 | 29
Not completed — Lost to Follow-up | 17 | 11
Not completed — Withdrawal by Subject | 3 | 0
Not completed — Death | 22 | 16
Not completed — Other | 1 | 0
Not completed — Randomized but Not Treated | 1 | 2

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) analysis set consisted of all participants who were randomized and treated in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Sirukumab + SOC | Placebo + SOC | Total
Number analyzed (Participants) | 139 | 70 | 209
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 94 | 48 | 142
  >=65 years | 45 | 22 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (12.91) | 57.8 (12.91) | 57.8 (12.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 25 | 66
  Male | 98 | 45 | 143
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 64 | 36 | 100
  Not Hispanic or Latino | 75 | 34 | 109
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 7 | 3 | 10
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 11 | 29
  White | 104 | 51 | 155
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 5 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  UNITED STATES | 139 | 70 | 209

OUTCOME MEASURES:

1. Primary Outcome: Time to Sustained Improvement of at Least 2 Categories on 6-point Ordinal Clinical Recovery Scale (CRS): Primary Analysis Set
Description: Time to sustained improvement is defined as an improvement of at least 2 categories relative to baseline on the 6-point ordinal clinical recovery scale sustained until Day 28. The 6-point ordinal CRS provides 6 mutually exclusive conditions ordered from best (score 1) to worst (score 6) corresponding to below categories, reflects the participant's worst situation on the day assessed. The ordinal clinical recovery scale categories are: not hospitalized, including participants on low level of oxygen (category 1); Hospitalization, not requiring supplemental oxygen (category 2); hospitalized, requiring low flow supplemental oxygen (category 3); hospitalized, on non-invasive pressure ventilation or high flow oxygen devices (category 4); hospitalized, on invasive mechanical ventilation (IMV) or extracorporeal membrane oxygenation (ECMO) (category 5); death (category 6). Higher scores indicated greater worsening.
Time Frame: Up to Day 28
Population: The Primary Analysis Set consisted of all participants in the Intent-to-Treat (ITT) analysis set (which consisted of all participants who were randomized and treated in the study) with confirmed critical COVID-19 disease defined as score of 4 or 5 on the ordinal CRS at baseline.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sirukumab + SOC | Placebo + SOC
Number analyzed (Participants) | 72 | 40
Days | 17.00 [13.00 to NA] — NA stands for data Not available as indicates upper limit of 95% CI was not estimable due to less number of events. | 23.00 [13.00 to NA] — NA stands for data Not available as indicates upper limit of 95% CI was not estimable due to less number of events.

2. Secondary Outcome: Percentage of Participants With an Improvement of At Least 2 Categories Compared to Baseline on 6-point Ordinal CRS
Description: Percentage of participants with an improvement of at least 2 Categories compared to baseline on 6-point ordinal CRS were reported. The 6-point ordinal CRS provides 6 mutually exclusive conditions ordered from best (score 1) to worst (score 6) corresponding to below categories, reflects the participant's worst situation on the day assessed. The ordinal clinical recovery scale categories are: not hospitalized, including participants on low level of oxygen (category 1); Hospitalization, not requiring supplemental oxygen (category 2); hospitalized, requiring low flow supplemental oxygen (category 3); hospitalized, on non-invasive pressure ventilation or high flow oxygen devices (category 4); hospitalized, on invasive mechanical ventilation (IMV) or extracorporeal membrane oxygenation (ECMO) (category 5); death (category 6). Higher scores indicated greater worsening.
Time Frame: Day 28
Population: The Primary Analysis Set consisted of all participants in the ITT analysis set with confirmed critical COVID-19 disease defined as score of 4 or 5 on the ordinal CRS at baseline. Here, 'N' (Number of participants analyzed) included all participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Sirukumab + SOC | Placebo + SOC
Number analyzed (Participants) | 69 | 40
Percentage of Participants | 59.4 | 55.0

3. Secondary Outcome: Percentage of Participants With All-cause Mortality Up to 28 Days
Description: Percentage of participants with all-cause mortality up to 28 days were reported. All-cause mortality included all deaths of participants due to any cause.
Time Frame: Up to 28 days
Population: as for outcome 2
Measure: Number; unit: Percentage of Participants
Arm/Group | Sirukumab + SOC | Placebo + SOC
Number analyzed (Participants) | 69 | 40
Percentage of Participants | 24.6 | 30.0

4. Secondary Outcome: Time to Sustained Improvement of at Least 2 Categories on 6-point Ordinal CRS: Intent-to-Treat (ITT) Set
Description: Time to sustained improvement is defined as an improvement of at least 2 categories relative to baseline on the 6-point ordinal clinical recovery scale, sustained until Day 28. The 6-point ordinal CRS provides 6 mutually exclusive conditions ordered from best (score 1) to worst (score 6) corresponding to below categories, reflects the participant's worst situation on the day assessed. The ordinal clinical recovery scale categories are: not hospitalized, including participants on low level of oxygen (category 1); Hospitalization, not requiring supplemental oxygen (category 2); hospitalized, requiring low flow supplemental oxygen (category 3); hospitalized, on non-invasive pressure ventilation or high flow oxygen devices (category 4); hospitalized, on invasive mechanical ventilation (IMV) or extracorporeal membrane oxygenation (ECMO) (category 5); death (category 6). Higher scores indicated greater worsening.
Time Frame: Up to Day 28
Population: The ITT analysis set consisted of all participants who were randomized and treated in the study.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Sirukumab + SOC | Placebo + SOC
Number analyzed (Participants) | 139 | 70
Days | 9.00 [7.00 to 10.00] | 10.00 [8.00 to 17.00]

5. Secondary Outcome: Percentage of Participants With an Improvement of at Least 2 Categories Compared to Baseline on 6-point Ordinal CRS: ITT Set
Description: as for outcome 2
Time Frame: Day 28
Population: The ITT analysis set consisted of all participants who were randomized and treated in the study. Here, 'N' (Number of participants analyzed) included all participants evaluable for this outcome measure. There were 3 participants in the 'Sirukumab + SOC arm' who discontinued the trial before Day 28 and thus were not evaluable for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Sirukumab + SOC | Placebo + SOC
Number analyzed (Participants) | 136 | 70
Percentage of Participants | 77.9 | 70.0

6. Secondary Outcome: Percentage of Participants With All-cause Mortality: ITT Set
Description: Percentage of participants with all-cause mortality were reported. All-cause mortality included all deaths of participants due to any cause.
Time Frame: Day 28
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Sirukumab + SOC | Placebo + SOC
Number analyzed (Participants) | 136 | 70
Percentage of Participants | 13.2 | 18.6

7. Secondary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) (Treatment Phase)
Description: Percentage of participants with SAEs were reported. SAE is any AE that results in: death, persistent or significant disability/incapacity, requires inpatient hospitalization or prolongation of existing hospitalization, is life-threatening experience, is a congenital anomaly/birth defect and may jeopardize participant and/or may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Up to Day 28
Population: The All Subjects treated analysis set consisted of all participants who received the study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Sirukumab + SOC | Placebo + SOC
Number analyzed (Participants) | 139 | 70
Percentage of Participants | 25.2 | 31.4

8. Secondary Outcome: Percentage of Participants With Related Adverse Events (AEs)
Description: Percentage of participants with related AEs were reported. An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study.
Time Frame: Up to Day 28
Population: The All Subjects Treated analysis set consisted of all participants who received the study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Sirukumab + SOC | Placebo + SOC
Number analyzed (Participants) | 139 | 70
Percentage of Participants | 11.5 | 7.1

9. Secondary Outcome: Percentage of Participants With Severe or Life-threatening, Bacterial, Invasive Fungal, Viral or Opportunistic Infections
Description: Percentage of participants with severe or Life-threatening, bacterial, invasive fungal, viral or opportunistic infections were reported.
Time Frame: Up to Day 28
Population: The All Subjects treated analysis set consisted of all participants who received the study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Sirukumab + SOC | Placebo + SOC
Number analyzed (Participants) | 139 | 70
Percentage of Participants | 11.5 | 11.4

10. Secondary Outcome: Percentage of Participants With Grade 3 and 4 Neutropenia and Lymphocytopenia
Description: Percentage of participants with Grade 3 and 4 neutropenia and lymphocytopenia were reported. The laboratory abnormalities were determined as per division of microbiology and infectious diseases (DMID) adult toxicity as Grade 1: mild (transient or mild discomfort [less than {<} 48 hours]; no medical intervention/therapy required); Grade 2: moderate (mild to moderate limitation in activity - some assistance may be needed; no or minimal medical intervention/therapy required); Grade 3: severe (severe marked limitation in activity, some assistance usually required; medical intervention/therapy required, hospitalizations possible); Grade 4: life-threatening (extreme limitation in activity, significant assistance required; significant medical intervention/therapy required, hospitalization or hospice care probable).
Time Frame: Up to Day 28
Population: The All Subjects Treated analysis set consists of all participants who received the study drug. Here, 'N' (Number of participants analyzed) included all participants evaluable for this outcome measure. Here, 'n' (number analyzed) is defined as participants analyzed for specified categories.
Measure: Number; unit: Percentage of Participants
Arm/Group | Sirukumab + SOC | Placebo + SOC
Number analyzed (Participants) | 137 | 69
Percentage of Participants
  Neutropenia: Grade 3: number analyzed (Participants) | 136 | 69
  Neutropenia: Grade 3 | 0 | 0
  Neutropenia: Grade 4: number analyzed (Participants) | 136 | 69
  Neutropenia: Grade 4 | 0.7 | 0
  Lymphocytopenia: Grade 3 | 6.6 | 7.2
  Lymphocytopenia: Grade 4 | 6.6 | 10.1

11. Secondary Outcome: Percentage of Participants With Increased Alanine Transaminase (ALT) Greater Than or Equal to (>=)3*Upper Limit Normal (ULN) Combined With Increased Bilirubin Greater Than (>)2*ULN
Description: Percentage of participants with increased ALT >=3*ULN combined with increased bilirubin >2*ULN were reported.
Time Frame: Up to Day 28
Population: The All Subjects Treated analysis set consists of all participants who received the study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Sirukumab + SOC | Placebo + SOC
Number analyzed (Participants) | 139 | 70
Percentage of Participants | 2.2 | 1.4

12. Secondary Outcome: Time to Sustained Improvement of at Least 1 Category on 6-point Ordinal CRS: Primary Analysis Set
Description: Time to sustained improvement is defined as an improvement of at least 1 category relative to baseline on the 6-point ordinal clinical recovery scale, sustained until Day 28. The 6-point ordinal CRS provides 6 mutually exclusive conditions ordered from best (score 1) to worst (score 6) corresponding to below categories, reflects the participant's worst situation on the day assessed. The ordinal clinical recovery scale categories are: not hospitalized, including participants on low level of oxygen (category 1); Hospitalization, not requiring supplemental oxygen (category 2); hospitalized, requiring low flow supplemental oxygen (category 3); hospitalized, on non-invasive pressure ventilation or high flow oxygen devices (category 4); hospitalized, on invasive mechanical ventilation (IMV) or extracorporeal membrane oxygenation (ECMO) (category 5); death (category 6). Higher scores indicated greater worsening.
Time Frame: Up to Day 28
Population: The Primary Analysis Set consisted of all participants in the ITT analysis set with confirmed critical COVID-19 disease defined as score of 4 or 5 on the ordinal CRS at baseline.
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | Sirukumab + SOC | Placebo + SOC
Number analyzed (Participants) | 72 | 40
Days | 9.00 [7.00 to 21.00] | 15.50 [8.00 to NA] — NA stands for data Not available, indicates upper limit of 90% CI was not estimable due to less number of events.

13. Secondary Outcome: Time to Sustained Improvement of at Least 1 Category on 6-point Ordinal CRS: ITT Set
Description: as for outcome 12
Time Frame: Up to Day 28
Population: The ITT analysis set consisted of all participants who were randomized and treated in the study.
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | Sirukumab + SOC | Placebo + SOC
Number analyzed (Participants) | 139 | 70
Days | 7.00 [6.00 to 8.00] | 7.00 [6.00 to 9.00]

14. Secondary Outcome: Percentage of Participants With an Improvement of at Least 1 Category Compared to Baseline on 6-point Ordinal CRS: Primary Analysis Set
Description: The 6-point ordinal CRS provides 6 mutually exclusive conditions ordered from best (score 1) to worst (score 6), reflects the participant's worst situation on the day assessed. The ordinal clinical recovery scale categories are: (category 1) not hospitalized, including participants on low level of oxygen; Hospitalization, not requiring supplemental oxygen (category 2); hospitalized, requiring low flow supplemental oxygen (category 3); hospitalized, on non-invasive pressure ventilation or high flow oxygen devices (category 4); hospitalized, on invasive mechanical ventilation (IMV) or extracorporeal membrane oxygenation (ECMO) (category 5); death (category 6). Higher scores indicated greater worsening.
Time Frame: Day 28
Population: The Primary Analysis Set consisted of all participants in the ITT analysis set with confirmed critical COVID-19 disease defined as score of 4 or 5 on the ordinal CRS at baseline. Here, 'N' (Number of participants analyzed) included all participants evaluable for this outcome measure. There were 3 participants in the 'Sirukumab + SOC arm' who discontinued the trial before Day 28 and thus were not evaluable for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Sirukumab + SOC | Placebo + SOC
Number analyzed (Participants) | 69 | 40
Percentage of Participants | 62.3 | 57.5

15. Secondary Outcome: Percentage of Participants With an Improvement of at Least 1 Category on 6-point Ordinal CRS: ITT Set
Description: The 6-point ordinal CRS provides 6 mutually exclusive conditions ordered from best (score 1) to worst (score 6) corresponding to below categories, reflects the participant's worst situation on the day assessed. The ordinal clinical recovery scale categories are: not hospitalized, including participants on low level of oxygen (category 1); Hospitalization, not requiring supplemental oxygen (category 2); hospitalized, requiring low flow supplemental oxygen (category 3); hospitalized, on non-invasive pressure ventilation or high flow oxygen devices (category 4); hospitalized, on invasive mechanical ventilation (IMV) or extracorporeal membrane oxygenation (ECMO) (category 5); death (category 6). Higher scores indicated greater worsening
Time Frame: Day 28
Population: as for outcome 5
Measure: Number; unit: Percentage of Participants
Arm/Group | Sirukumab + SOC | Placebo + SOC
Number analyzed (Participants) | 136 | 70
Percentage of Participants | 80.1 | 74.3

16. Secondary Outcome: Time From Study Intervention Administration to End of Oxygen Supplementation
Description: Time from study intervention administration to end of oxygen supplementation was reported.
Time Frame: Up to Day 28
Population: The ITT analysis set consisted of all participants who were randomized and treated in the study.
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | Sirukumab + SOC | Placebo + SOC
Number analyzed (Participants) | 139 | 70
Days | 24.0 [10.00 to NA] — NA indicates data not available as upper limit of 90% CI was not estimable due to less number of events. | 20.00 [9.00 to NA] — NA indicates data not available as upper limit of 90% CI was not estimable due to less number of events.

17. Secondary Outcome: Time From Study Intervention Administration to Hospital Discharge Among the Surviving Participants
Description: Time from study intervention administration to hospital discharge among the surviving participants was reported.
Time Frame: Up to Day 28
Population: The ITT population restricted to participants surviving up to Day 28.
Measure: Median (90% Confidence Interval); unit: Days
Arm/Group | Sirukumab + SOC | Placebo + SOC
Number analyzed (Participants) | 118 | 57
Days | 8.00 [7.00 to 9.00] | 9.00 [7.00 to 10.00]

18. Secondary Outcome: Total Length of Hospitalization Among the Surviving Participants
Description: Total length of hospitalization, defined as total duration of hospital stay, among the surviving participants was reported.
Time Frame: Up to Day 28
Population: The ITT population restricted to participants surviving up to Day 28.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Sirukumab + SOC | Placebo + SOC
Number analyzed (Participants) | 118 | 57
Days | 10.42 (8.274) | 11.19 (8.370)

19. Secondary Outcome: Number of Ventilation Free Days
Description: Number of ventilation free days in participants on invasive mechanical ventilation (IVM)/extracorporeal membrane oxygenation (ECMO) at baseline was reported.
Time Frame: Up to Day 28
Population: The Primary Analysis Set restricted to participants who were on IVM/ECMO at baseline. Here, 'N' (Number of participants analyzed) included all participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Sirukumab + SOC | Placebo + SOC
Number analyzed (Participants) | 11 | 8
Days | 13.82 (11.062) | 6.63 (9.546)

20. Secondary Outcome: Percentage of Participants With Clinical Status as Assessed by 6-point Ordinal CRS: Primary Analysis Set
Description: Percentage of participants with clinical status as assessed by 6-point Ordinal CRS were reported. The 6-point ordinal CRS provides 6 mutually exclusive conditions ordered from best (score 1) to worst (score 6) corresponding to below categories, reflects the participant's worst situation on the day assessed. The ordinal clinical recovery scale categories are: Not hospitalized, not requiring supplemental oxygen (category 1.1); Not hospitalized, requiring supplemental oxygen (category 1.2); Hospitalization, not requiring supplemental oxygen (category 2); hospitalized, requiring low flow supplemental oxygen (category 3); hospitalized, on non-invasive pressure ventilation or high flow oxygen devices (category 4); hospitalized, on invasive mechanical ventilation (IMV) or extracorporeal membrane oxygenation (ECMO) (category 5); death (category 6). Higher scores indicated greater worsening.
Time Frame: On Day 7, 14, 21, 28
Population: The Primary Analysis Set consisted of all participants in the ITT set with confirmed critical COVID-19 disease defined as score of 4 or 5 on ordinal CRS at baseline. Here 'N' (number of participants analyzed) included all participants evaluable for this outcome measure. Here, 'n' (number analyzed) is defined as participants analyzed for specified categories at specified timepoints.
Measure: Number; unit: Percentage of Participants
Arm/Group | Sirukumab + SOC | Placebo + SOC
Number analyzed (Participants) | 71 | 40
Percentage of Participants
  Day 7: Category 1.1 | 7.0 | 5.0
  Day 7: Category 1.2 | 4.2 | 2.5
  Day 7: Category 2 | 4.2 | 0
  Day 7: Category 3 | 22.5 | 25.0
  Day 7: Category 4 | 33.8 | 32.5
  Day 7: Category 5 | 25.4 | 35.0
  Day 7: Category 6 | 2.8 | 0
  Day 14: Category 1.1: number analyzed (Participants) | 69 | 40
  Day 14: Category 1.1 | 20.3 | 17.5
  Day 14: Category 1.2: number analyzed (Participants) | 69 | 40
  Day 14: Category 1.2 | 20.3 | 15.0
  Day 14: Category 2: number analyzed (Participants) | 69 | 40
  Day 14: Category 2 | 1.4 | 2.5
  Day 14: Category 3: number analyzed (Participants) | 69 | 40
  Day 14: Category 3 | 13.0 | 15.0
  Day 14: Category 4: number analyzed (Participants) | 69 | 40
  Day 14: Category 4 | 13.0 | 10.0
  Day 14: Category 5: number analyzed (Participants) | 69 | 40
  Day 14: Category 5 | 20.3 | 27.5
  Day 14: Category 6: number analyzed (Participants) | 69 | 40
  Day 14: Category 6 | 11.6 | 12.5
  Day 21: Category 1.1: number analyzed (Participants) | 69 | 40
  Day 21: Category 1.1 | 23.2 | 20.0
  Day 21: Category 1.2: number analyzed (Participants) | 69 | 40
  Day 21: Category 1.2 | 26.1 | 22.5
  Day 21: Category 2: number analyzed (Participants) | 69 | 40
  Day 21: Category 2 | 1.4 | 7.5
  Day 21: Category 3: number analyzed (Participants) | 69 | 40
  Day 21: Category 3 | 10.1 | 5.0
  Day 21: Category 4: number analyzed (Participants) | 69 | 40
  Day 21: Category 4 | 7.2 | 5.0
  Day 21: Category 5: number analyzed (Participants) | 69 | 40
  Day 21: Category 5 | 17.4 | 20.0
  Day 21: Category 6: number analyzed (Participants) | 69 | 40
  Day 21: Category 6 | 14.5 | 20.0
  Day 28: Category 1.1: number analyzed (Participants) | 69 | 40
  Day 28: Category 1.1 | 29.0 | 25.0
  Day 28: Category 1.2: number analyzed (Participants) | 69 | 40
  Day 28: Category 1.2 | 27.5 | 25.0
  Day 28: Category 2: number analyzed (Participants) | 69 | 40
  Day 28: Category 2 | 0 | 5.0
  Day 28: Category 3: number analyzed (Participants) | 69 | 40
  Day 28: Category 3 | 5.8 | 2.5
  Day 28: Category 4: number analyzed (Participants) | 69 | 40
  Day 28: Category 4 | 4.3 | 0
  Day 28: Category 5: number analyzed (Participants) | 69 | 40
  Day 28: Category 5 | 8.7 | 12.5
  Day 28: Category 6: number analyzed (Participants) | 69 | 40
  Day 28: Category 6 | 24.6 | 30.0

21. Secondary Outcome: Percentage of Participants With Clinical Status as Assessed by 6-point Ordinal CRS: ITT Set
Description: Percentage of participants with clinical status as assessed by 6-point Ordinal CRS (ITT Set) were reported. The 6-point ordinal CRS provides 6 mutually exclusive conditions ordered from best (score 1) to worst (score 6) corresponding to below categories, reflects the participant's worst situation on the day assessed. The ordinal clinical recovery scale categories are: Not hospitalized, not requiring supplemental oxygen (category 1.1); Not hospitalized, requiring supplemental oxygen (category 1.2); Hospitalization, not requiring supplemental oxygen (category 2); hospitalized, requiring low flow supplemental oxygen (category 3); hospitalized, on non-invasive pressure ventilation or high flow oxygen devices (category 4); hospitalized, on invasive mechanical ventilation (IMV) or extracorporeal membrane oxygenation (ECMO) (category 5); death (category 6). Higher scores indicated greater worsening.
Time Frame: On Days 7, 14, 21, 28
Population: The ITT analysis set consisted of all participants who were randomized and treated in the study. Here 'N' (number of participants analyzed) included all participants evaluable for this outcome measure. Here, 'n' (number analyzed) is defined as participants analyzed for specified categories at specified timepoints.
Measure: Number; unit: Percentage of Participants
Arm/Group | Sirukumab + SOC | Placebo + SOC
Number analyzed (Participants) | 138 | 70
Percentage of Participants
  Day 7: Category 1.1 | 31.9 | 30.0
  Day 7: Category 1.2 | 8.7 | 5.7
  Day 7: Category 2 | 5.1 | 4.3
  Day 7: Category 3 | 20.3 | 20.0
  Day 7: Category 4 | 18.8 | 18.6
  Day 7: Category 5 | 13.8 | 21.4
  Day 7: Category 6 | 1.4 | 0
  Day 14: Category 1.1: number analyzed (Participants) | 136 | 70
  Day 14: Category 1.1 | 44.1 | 42.9
  Day 14: Category 1.2: number analyzed (Participants) | 136 | 70
  Day 14: Category 1.2 | 24.3 | 17.1
  Day 14: Category 2: number analyzed (Participants) | 136 | 70
  Day 14: Category 2 | 0.7 | 1.4
  Day 14: Category 3: number analyzed (Participants) | 136 | 70
  Day 14: Category 3 | 6.6 | 8.6
  Day 14: Category 4: number analyzed (Participants) | 136 | 70
  Day 14: Category 4 | 7.4 | 5.7
  Day 14: Category 5: number analyzed (Participants) | 136 | 70
  Day 14: Category 5 | 10.3 | 15.7
  Day 14: Category 6: number analyzed (Participants) | 136 | 70
  Day 14: Category 6 | 6.6 | 8.6
  Day 21: Category 1.1: number analyzed (Participants) | 136 | 70
  Day 21: Category 1.1 | 45.6 | 44.3
  Day 21: Category 1.2: number analyzed (Participants) | 136 | 70
  Day 21: Category 1.2 | 27.9 | 21.4
  Day 21: Category 2: number analyzed (Participants) | 136 | 70
  Day 21: Category 2 | 0.7 | 4.3
  Day 21: Category 3: number analyzed (Participants) | 136 | 70
  Day 21: Category 3 | 5.1 | 2.9
  Day 21: Category 4: number analyzed (Participants) | 136 | 70
  Day 21: Category 4 | 3.7 | 2.9
  Day 21: Category 5: number analyzed (Participants) | 136 | 70
  Day 21: Category 5 | 8.8 | 11.4
  Day 21: Category 6: number analyzed (Participants) | 136 | 70
  Day 21: Category 6 | 8.1 | 12.9
  Day 28: Category 1.1: number analyzed (Participants) | 136 | 70
  Day 28: Category 1.1 | 48.5 | 47.1
  Day 28: Category 1.2: number analyzed (Participants) | 136 | 70
  Day 28: Category 1.2 | 28.7 | 22.9
  Day 28: Category 2: number analyzed (Participants) | 136 | 70
  Day 28: Category 2 | 0 | 2.9
  Day 28: Category 3: number analyzed (Participants) | 136 | 70
  Day 28: Category 3 | 2.9 | 1.4
  Day 28: Category 4: number analyzed (Participants) | 136 | 70
  Day 28: Category 4 | 2.2 | 0
  Day 28: Category 5: number analyzed (Participants) | 136 | 70
  Day 28: Category 5 | 4.4 | 7.1
  Day 28: Category 6: number analyzed (Participants) | 136 | 70
  Day 28: Category 6 | 13.2 | 18.6

22. Secondary Outcome: Total Time on Invasive Mechanical Ventilation
Description: Total time on invasive mechanical ventilation in participants who were on invasive mechanical ventilation at baseline was reported.
Time Frame: Up to Day 28
Population: The Primary Analysis Set restricted to participants who were on invasive mechanical ventilation at baseline. Here 'N' (number of participants analyzed) included all participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Sirukumab + SOC | Placebo + SOC
Number analyzed (Participants) | 11 | 8
Days | 14.18 (11.062) | 21.37 (9.546)

23. Secondary Outcome: Percentage of Participants With a Worse Category Relative to Baseline on the 6-point Ordinal CRS
Description: Percentage of participants with a worse category relative to baseline on the 6-point ordinal CRS for at least one of the daily assessment during the reporting period Day 5 and Day 28 were reported. he 6-point ordinal CRS provides 6 mutually exclusive conditions ordered from best (score 1) to worst (score 6) corresponding to below categories, reflects the participant's worst situation on the day assessed. The ordinal clinical recovery scale categories are: not hospitalized, including participants on low level of oxygen (category 1); Hospitalization, not requiring supplemental oxygen (category 2); hospitalized, requiring low flow supplemental oxygen (category 3); hospitalized, on non-invasive pressure ventilation or high flow oxygen devices (category 4); hospitalized, on invasive mechanical ventilation (IMV) or extracorporeal membrane oxygenation (ECMO) (category 5); death (category 6). Higher scores indicated greater worsening.
Time Frame: From Day 5 up to Day 28
Population: The ITT analysis set consisted of all participants who were randomized and treated in the study. Here 'N' (number of participants analyzed) included all participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Sirukumab + SOC | Placebo + SOC
Number analyzed (Participants) | 136 | 70
Percentage of Participants | 25.0 | 31.4

24. Secondary Outcome: Percentage of Participants With Extracorporeal Membrane Oxygenation (ECMO) Over Time
Description: Percentage of participants with ECMO over time were reported.
Time Frame: From Day 1 up to Day 28
Population: The ITT population restricted to participants who were on ECMO at baseline.
Measure: Number; unit: Percentage of Participants
Arm/Group | Sirukumab + SOC | Placebo + SOC
Number analyzed (Participants) | 2 | 3
Percentage of Participants
  Day 1 | 100.0 | 100.0
  Day 2 | 0 | 33.3
  Day 3 | 0 | 0
  Day 4 | 0 | 0
  Day 5 | 0 | 0
  Day 6 | 0 | 0
  Day 7 | 0 | 0
  Day 8 | 0 | 0
  Day 9 | 0 | 0
  Day 10 | 0 | 0
  Day 11 | 0 | 0
  Day 12 | 0 | 0
  Day 13 | 0 | 0
  Day 14 | 0 | 0
  Day 15 | 0 | 0
  Day 16 | 0 | 0
  Day 17 | 0 | 0
  Day 18 | 0 | 0
  Day 19 | 0 | 0
  Day 20 | 0 | 0
  Day 21 | 0 | 0
  Day 22 | 0 | 0
  Day 23 | 0 | 0
  Day 24 | 0 | 0
  Day 25 | 0 | 0
  Day 26 | 0 | 0
  Day 27 | 0 | 0
  Day 28 | 0 | 0

25. Secondary Outcome: Total Time on ECMO
Description: Total time for participants on ECMO was reported.
Time Frame: Up to Day 28
Population: The ITT set restricted to participants who were on ECMO at baseline.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Sirukumab + SOC | Placebo + SOC
Number analyzed (Participants) | 2 | 3
Days | 1.0 (0) | 1.3 (0.58)

26. Secondary Outcome: Percentage of Alive Participants at Day 28, Week 8, and Week 16
Description: Percentage of alive participants at Day 28, Week 8, and Week 16 were reported. For this outcome measure, at Week 8, data was not collected for participants due to pandemic situation.
Time Frame: On Day 28, Week 8 and Week 16
Population: The ITT analysis set consisted of all participants who were randomized and treated in the study. Here 'N' (number of participants analyzed) included all participants evaluable for this outcome measure. Here, 'n' (number analyzed) is defined as participants analyzed for specified timepoints.
Measure: Number; unit: Percentage of Participants
Arm/Group | Sirukumab + SOC | Placebo + SOC
Number analyzed (Participants) | 136 | 70
Percentage of Participants
  Day 28 | 86.8 | 81.4
  Week 8: number analyzed (Participants) | 0 | 0
  Week 16: number analyzed (Participants) | 118 | 59
  Week 16 | 81.3 | 72.9

27. Secondary Outcome: Percentage of Alive Participants That Required Readmission at Week 8, and Week 16
Description: Percentage of alive participants that required readmission at Week 8, and Week 16 were reported. For this outcome measure, at Week 8 and Week 16, data was not collected for participants due to pandemic situation.
Time Frame: Week 8 and Week 16
Population: The ITT analysis set consisted of all participants who were randomized and treated in the study.
Measure: Number; unit: Percentage of Participants
Arm/Group | Sirukumab + SOC | Placebo + SOC
Number analyzed (Participants) | 139 | 70

28. Secondary Outcome: Percentage of Participants With SAEs (Follow-up Phase)
Description: as for outcome 7
Time Frame: From Week 4 up to Week 16
Population: The All Subjects Treated analysis set consists of all participants who received the study drug. Here, 'N' (Number of participants analyzed) included all participants evaluable for this outcome measure.
Measure: Number; unit: Percentage of Participants
Arm/Group | Sirukumab + SOC | Placebo + SOC
Number analyzed (Participants) | 118 | 57
Percentage of Participants | 5.9 | 5.3

ADVERSE EVENTS:
Time Frame: Treatment phase: Weeks 0-4; Follow-up phase: Weeks 4-16
Description: The All Subjects Treated analysis set consisted of all participants who received the study drug. The number of participants at risk in placebo arm in follow-up phase were 59 participants, however, the data for 2 participants in placebo arms were not collected due to pandemic situation, and were excluded from the analysis. Therefore, here number of participants at risk are 57 participants.
Groups:
- Sirukumab + Standard of Care (SOC): Treatment Phase: Hospitalized participants with confirmed coronavirus disease-2019 (COVID-19) received intravenous (IV) single dose infusion of sirukumab (5 milligrams per kilogram [mg/kg]) on Day 1 along with SOC treatment per the discretion of the Investigator.
- Sirukumab + SOC: Follow-up Phase: Hospitalized participants with confirmed COVID-19 received IV single dose infusion of sirukumab 5 mg/kg on Day 1 along with SOC treatment per the discretion of the Investigator.
- Placebo + SOC: Treatment Phase; Placebo + SOC: Follow-up Phase: Hospitalized participants with confirmed COVID-19 disease received IV single dose infusion of placebo on Day 1 along with SOC treatment per the discretion of the Investigator.
Arm/Group | Sirukumab + Standard of Care (SOC): Treatment Phase | Sirukumab + SOC: Follow-up Phase | Placebo + SOC: Treatment Phase | Placebo + SOC: Follow-up Phase
All-Cause Mortality (participants affected / at risk) | 18/139 | 4/118 | 13/70 | 3/57
Serious Adverse Events (participants affected / at risk) | 35/139 | 7/118 | 22/70 | 3/57
Other Adverse Events (participants affected / at risk) | 24/139 | 1/118 | 16/70 | 1/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sirukumab + Standard of Care (SOC): Treatment Phase (N=139) | Sirukumab + SOC: Follow-up Phase (N=118) | Placebo + SOC: Treatment Phase (N=70) | Placebo + SOC: Follow-up Phase (N=57)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Blood Loss Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Disseminated Intravascular Coagulation (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0
Acute Left Ventricular Failure (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac Arrest (Cardiac disorders) | 3 | 1 | 6 | 0
Cardio-Respiratory Arrest (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiogenic Shock (Cardiac disorders) | 2 | 0 | 0 | 0
Myocardial Ischaemia (Cardiac disorders) | 0 | 1 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Lower Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mallory-Weiss Syndrome (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Mouth Haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Retroperitoneal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Multiple Organ Dysfunction Syndrome (General disorders) | 0 | 0 | 2 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 1
Bacterial Sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Covid-19 (Infections and infestations) | 3 | 0 | 1 | 0
Covid-19 Pneumonia (Infections and infestations) | 0 | 1 | 1 | 0
Enterobacter Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Enterococcal Bacteraemia (Infections and infestations) | 0 | 1 | 0 | 0
Hiv Infection (Infections and infestations) | 1 | 0 | 0 | 0
Klebsiella Infection (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 0
Septic Shock (Infections and infestations) | 2 | 0 | 2 | 0
Staphylococcal Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Streptococcal Bacteraemia (Infections and infestations) | 1 | 0 | 0 | 0
Viral Sepsis (Infections and infestations) | 2 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 0 | 0
Glomerular Filtration Rate Decreased (Investigations) | 0 | 0 | 1 | 0
Hepatic Enzyme Increased (Investigations) | 0 | 0 | 1 | 0
Transaminases Increased (Investigations) | 1 | 0 | 0 | 0
Urine Analysis Abnormal (Investigations) | 0 | 0 | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 1 | 0
Embolic Stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Haemorrhage Intracranial (Nervous system disorders) | 0 | 0 | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 1 | 1 | 4 | 0
Oliguria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal Impairment (Renal and urinary disorders) | 2 | 0 | 1 | 0
Acute Respiratory Distress Syndrome (Respiratory, thoracic and mediastinal disorders) | 12 | 1 | 5 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 6 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 6 | 0 | 2 | 0
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumomediastinum (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 3 | 0
Pneumothorax Spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 6 | 0
Subcutaneous Emphysema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Haemodialysis (Surgical and medical procedures) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 2 | 0 | 0 | 0
Orthostatic Hypotension (Vascular disorders) | 1 | 1 | 0 | 0
Shock (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sirukumab + Standard of Care (SOC): Treatment Phase (N=139) | Sirukumab + SOC: Follow-up Phase (N=118) | Placebo + SOC: Treatment Phase (N=70) | Placebo + SOC: Follow-up Phase (N=57)
Leukocytosis (Blood and lymphatic system disorders) | 8 | 1 | 6 | 0
Alanine Aminotransferase Increased (Investigations) | 7 | 0 | 2 | 0
Transaminases Increased (Investigations) | 8 | 0 | 2 | 0
Troponin Increased (Investigations) | 1 | 0 | 4 | 0
Acute Kidney Injury (Renal and urinary disorders) | 4 | 0 | 5 | 1
Hypotension (Vascular disorders) | 5 | 0 | 5 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. Expedited reviews will be arranged for abstracts, poster presentations, or other materials. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2021-02-17): https://cdn.clinicaltrials.gov/large-docs/61/NCT04380961/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-28): https://cdn.clinicaltrials.gov/large-docs/61/NCT04380961/SAP_001.pdf